CLINICAL TRIAL: NCT05530772
Title: Immediate Endoscopic Necrosectomy vs. On-demand Necroectomy in Infected Walled-off Pancreatic Necrosis
Brief Title: Immediate vs. On-demand Endoscopic Necrosectomy in Infected Walled-off Pancreatic Necrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tehran (Other)
Responsible Party: Principal Investigator, Mehdi Mohamadnejad, Associate professor of medicine, University of Tehran
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DDRI.1401.008
Record Dates: First submitted 2022-09-02; First posted 2022-09-07 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Pancreatitis, Acute Necrotizing
MeSH Terms: conditions — Pancreatitis, Acute Necrotizing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Immediate endoscopic Necrosectomy (Experimental): The subject will have endoscopic necrosectomy at the time of the EUS-guided transmural stent placement.
  The necrotic collection is identified with endoscopic ultrasonography (EUS). Transmural placement of stent under EUS guidance is performed. The type of stent is at the discretion of endoscopist. It could be either lumen apposing metallic stent or double pigtail plastic stent. Immediately after stent placement, the cystoenterostomy track is dilated with a 15 mm through the scope (TTS) balloon. Then, direct endoscopic necrosectomy is performed with CO2 insufflation. The duration of necrosectomy will be 30 to 90 minutes. If complete clearance of the cavity is achieved before 30 minutes, the duration of necrosectomy may be less than 30 minutes in the given session. Also, if any complication occurs during necrosectomy, appropriate management will be done, and the procedure may be concluded earlier.
  Interventions: Device: Endoscopic necrosectomy
- On-demand endoscopic necrosectomy (Active Comparator): The subject will have EUS-guided transmural drainage of the necrotic collection The necrotic collection is identified with endoscopic ultrasonography (EUS). Transmural placement of stent under EUS guidance is performed. The type of stent is at the discretion of endoscopist. It could be either lumen apposing metallic stent or double pigtail plastic stent. In this group, endoscopic necrosectomy is not performed at the time of index procedure. Such patients may undergo endoscopic necrosectomy during follow up if clinically indicated.
  Interventions: Device: Endoscopic necrosectomy

INTERVENTIONS:
Device: Endoscopic necrosectomy — Initially, a tract is created between the stomach or duodenum with the walled-off pancreatic necrotic collection through placement of a stent. Then, the endosocpe is entered the necrotic cavity with CO2 insufflation, and the necrotic materials are removed with snare, grasper, or suctioning.

SUMMARY:
Acute pancreatitis is one of the most common diagnoses made in gastroenterology wards worldwide which causes a great deal of pain and expense along with fatal complications. Approximately, 10-20% of patients progress to necrotizing pancreatitis that result in significant morbidity and mortality. Initial conservative management may be feasible in necrotizing pancreatitis, however the majority of patients with infected necrosis or persistent symptoms will eventually require a drainage procedure. Drainage procedures for necrotizing pancreatitis include open surgery, minimally invasive surgery, percutaneous drainage, and endoscopic drainage. In the recent years, minimally invasive approaches have largely replaced open surgical necrosectomy. Endoscopic drainage of walled off pancreatic necrosis involves creation of a transmural fistula between the enteral lumen and WOPN cavity with stent placement under endoscopic ultrasound (EUS) guidance. Furthermore, direct endoscopic necrosectomy can be performed through the fistula track. The best timing for endoscopic necrosectomy is not yet defined. A recent retrospective study suggested that immediate necrosectomy after stent placement results in earlier resolution of WOPN with fewer sessions of endoscopic necrosectomy. The aim of this study is to compare immediate vs. on-demand endoscopic necrosectomy in patients with infected WOPN who undergo EUS-guided transmural drainage of WOPN.

DETAILED DESCRIPTION:
Acute pancreatitis is one of the most common diagnoses made in gastroenterology wards worldwide which causes a great deal of pain and expense along with fatal complications (1). The incidence of acute pancreatitis is trending upward in the United States with $2.6 billion annual health care costs (2). While most patients present with mild and interstitial form of pancreatitis, 10-20% of patients progress to necrotizing pancreatitis that result in significant morbidity and mortality (3). Initial conservative management may be feasible in necrotizing pancreatitis (4), however the majority of patients with infected necrosis or persistent symptoms will eventually require a drainage procedure (5). Drainage procedures for necrotizing pancreatitis include open surgery, minimally invasive surgery, percutaneous drainage, and endoscopic drainage. Drainage procedures are typically postponed for several weeks until the necrotic cavity becomes walled off which is called walled off pancreatic necrosis (WOPN).

In the recent years, minimally invasive approaches have largely replaced open surgical necrosectomy (6). Endoscopic drainage of walled off pancreatic necrosis involves creation of a transmural fistula between the enteral lumen and WOPN cavity with stent placement under endoscopic ultrasound (EUS) guidance. Furthermore, direct endoscopic necrosectomy can be performed through the fistula track. The best timing for endoscopic necrosectomy is not yet defined. A recent retrospective study suggested that immediate necrosectomy after stent placement results in earlier resolution of WOPN with fewer sessions of endoscopic necrosectomy (7).

The aim of this study is to compare immediate vs. on-demand endoscopic necrosectomy in patients with infected WOPN who undergo EUS-guided transmural drainage of WOPN.

Infected necrosis is diagnosed with one of the following criteria in patients with WOPN three weeks after onset of acute pancreatitis (8): A. Positive Gram's stain or culture from a fine-needle aspiration; B. the presence of gas within pancreatic and peripancreatic necrosis on contrast-enhanced CT scan; C. Presence of two inflammatory variables (temperature >38.5°C or elevated C-reactive protein levels or leukocyte counts) in the absence of another focus of infection (other than infected necrosis) ; D. Presence of persistent organ failure.

ELIGIBILITY:
Inclusion Criteria:

* Documented history of acute pancreatitis
* Necrotic collection with partial or complete wall diagnosed on CT or MRI
* Necrotic collection of any size with any number of loculations with more than 20% of solid/necrotic component
* Necrotic collection is accessible and amenable for EUS-guided drainage
* Age >= 18 years
* Suspected or confirmed infection in the necrotic collection
* The patient understands and accepts to sign the informed consent.

Exclusion Criteria:

* Irreversible coagulopathy with INR>1.5 or platelet counts <50,000
* Necrotic collection is not accessible for EUS-guided drainage
* Females who are pregnant
* Previous intervention (e,g, percutaneous drainage, or surgery) is performed for the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-09-12 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Clinical success rate | Three months
  Clinical success rate is compared between the two groups. Clinical success is defined as complete resolution of WOPN without residual fluid component along with resolution of symptoms three months after stent placement

SECONDARY OUTCOMES:
procedure-related adverse events | Three months
  Comparing procedure-related adverse events between the two groups. Adverse events including bleeding, perforation, secondary infection are compared.
Length of hospital stay | Three months
  Comparing length of hospital stay between the two groups. Total length of hospital stay is recorded and compared.
Number of necrosectomy sessions | Three months
  Comparing number of necrosectomy sessions between the two groups
Total duration of necrosectomies (in miniute) | Three months
  Comparing total duration of necrosectomies (in miniute) between the two groups. Total duration of necrosectomies (in miniute) in all necroectomy sessions is recorded and compared between the two groups.
Rate of new onset diabetes mellitus | Three months
  Comparing rate of new onset diabetes mellitus between the two groups
Mortality rate | Three months
  Comparing mortality rate between the two groups
Number of patients requiring surgery | Three months
  Comparing number of patients requiring surgery between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Alireza Delavari, MD, Study Chair — Chair, Digestive dieseases research institute, Tehran University of Medical Sciences
Locations (1):
- Digestive Diseases Research Institute, Shariati Hospital, North Kargar Ave.,, Tehran, Tehran Province, Iran

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared with other researchers for collaborative studies upon request from the principle investigator
Supporting Information: Study Protocol, CSR

REFERENCES:
- [Result] Lankisch PG, Apte M, Banks PA. Acute pancreatitis. Lancet. 2015 Jul 4;386(9988):85-96. doi: 10.1016/S0140-6736(14)60649-8. Epub 2015 Jan 21. PMID 25616312
- [Result] Peery AF, Crockett SD, Barritt AS, Dellon ES, Eluri S, Gangarosa LM, Jensen ET, Lund JL, Pasricha S, Runge T, Schmidt M, Shaheen NJ, Sandler RS. Burden of Gastrointestinal, Liver, and Pancreatic Diseases in the United States. Gastroenterology. 2015 Dec;149(7):1731-1741.e3. doi: 10.1053/j.gastro.2015.08.045. Epub 2015 Aug 29. PMID 26327134
- [Result] Baron TH, DiMaio CJ, Wang AY, Morgan KA. American Gastroenterological Association Clinical Practice Update: Management of Pancreatic Necrosis. Gastroenterology. 2020 Jan;158(1):67-75.e1. doi: 10.1053/j.gastro.2019.07.064. Epub 2019 Aug 31. PMID 31479658
- [Result] Mouli VP, Sreenivas V, Garg PK. Efficacy of conservative treatment, without necrosectomy, for infected pancreatic necrosis: a systematic review and meta-analysis. Gastroenterology. 2013 Feb;144(2):333-340.e2. doi: 10.1053/j.gastro.2012.10.004. Epub 2012 Oct 12. PMID 23063972
- [Result] Boxhoorn L, Voermans RP, Bouwense SA, Bruno MJ, Verdonk RC, Boermeester MA, van Santvoort HC, Besselink MG. Acute pancreatitis. Lancet. 2020 Sep 5;396(10252):726-734. doi: 10.1016/S0140-6736(20)31310-6. PMID 32891214
- [Result] van Santvoort HC, Besselink MG, Bakker OJ, Hofker HS, Boermeester MA, Dejong CH, van Goor H, Schaapherder AF, van Eijck CH, Bollen TL, van Ramshorst B, Nieuwenhuijs VB, Timmer R, Lameris JS, Kruyt PM, Manusama ER, van der Harst E, van der Schelling GP, Karsten T, Hesselink EJ, van Laarhoven CJ, Rosman C, Bosscha K, de Wit RJ, Houdijk AP, van Leeuwen MS, Buskens E, Gooszen HG; Dutch Pancreatitis Study Group. A step-up approach or open necrosectomy for necrotizing pancreatitis. N Engl J Med. 2010 Apr 22;362(16):1491-502. doi: 10.1056/NEJMoa0908821. PMID 20410514
- [Result] Yan L, Dargan A, Nieto J, Shariaha RZ, Binmoeller KF, Adler DG, DeSimone M, Berzin T, Swahney M, Draganov PV, Yang DJ, Diehl DL, Wang L, Ghulab A, Butt N, Siddiqui AA. Direct endoscopic necrosectomy at the time of transmural stent placement results in earlier resolution of complex walled-off pancreatic necrosis: Results from a large multicenter United States trial. Endosc Ultrasound. 2019 May-Jun;8(3):172-179. doi: 10.4103/eus.eus_108_17. PMID 29882517